CLINICAL TRIAL: NCT02493348
Title: A Study of the Effect of Rhythmic Sensory Stimulation on Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Allan Gordon, Director of Wasser Pain Management Centre, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSH REB 15-0140-E
Record Dates: First submitted 2015-07-02; First posted 2015-07-09 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Rhythmic Sensory Stimulation; Gamma Stimulation
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous 40 Hz Rhythmic Sensory Stimulation (Experimental): The intervention consists of Rhythmic Sensory Stimulation of a continuous sine wave single-frequency stimulation (40 Hz). The treatment prescription is 30 minutes daily 40 Hz Rhythmic Sensory Stimulation, 5 days per week, for five weeks of treatment, for a total of 25 sessions.
  Interventions: Device: Rhythmic Sensory Stimulation
- Intermittent Rhythmic Sensory Stimulation (Active Comparator): The stimulation consists of random and intermittent complex wave gamma-range RSS with peaks at 45 Hz and 95 Hz, for 30 minutes daily stimulation, 5 days per week, for a total of five weeks of treatment.
  Interventions: Device: Rhythmic Sensory Stimulation

INTERVENTIONS:
Device: Rhythmic Sensory Stimulation — Rhythmic Sensory Stimulation (RSS) can be delivered through sound devices. In this study, the stimuli will be delivered with a portable consumer device called Sound Oasis Vibroacoustic Therapy System (VTS) 1000 unit, which is a low-voltage consumer product device that has two built-in mid to high-frequency speakers and one built in low frequency (subwoofer-type) speaker. The low frequency sounds played by the subwoofer speaker is experienced as vibrotactile vibration. Although the Intervention of Interest in this study is the gamma-frequency acoustic-driven rhythmic sensory stimulation, the efficacy of the Sound Oasis VTS-1000 device to deliver this sound will also be observed.

SUMMARY:
Fibromyalgia is a chronic pain disorder associated with widespread pain that dramatically impacts patient's quality of life. The present research aims to determine the effectiveness of Rhythmic Sensory Stimulation with rhythmic gamma-frequency (30 - 120 Hz) acoustic-driven stimulation of mechanoreceptors in the body on the treatment of fibromyalgia. The proposed treatment involves 30 minutes of daily rhythmic vibroacoustic stimulation at gamma range, 5 days per week, for 5 weeks. Measures of pain severity, fibromyalgia symptoms, sleep quality, and depression, will be compared before and after treatment between the treatment and control groups. The results of the present study will help to better understand the effectiveness of Rhythmic Sensory Stimulation to the treatment of chronic pain disorders, such as fibromyalgia, and contribute to the development of future studies to investigate the neural driving effects of therapies based on Rhythmic Sensory Stimulation.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic pain disorder associated with widespread pain that dramatically impacts patients' quality of life. Its exact cause has not yet been identified, however, recent studies indicate that fibromyalgia is associated with a significant imbalance of the connectivity within brain networks associated with pain, decreased functional connectivity in the descending pain-modulating system, and increased activity in the pain matrix related to central sensitization. It has been suggested that treatments that stimulate or induce coherent neuronal activity, and synchronize dysregulated brain circuitry, have significant benefits in improving pain management and enhancing patients' quality of life.

An example of a non-invasive treatment that is thought to indirectly stimulate neuronal coherence is Rhythmic Sensory Stimulation (RSS) in gamma frequencies. RSS stimulates the mechanoreceptors in the body using gamma-frequency sounds (e.g., 40 Hz) by means of speakers in a chair. Previous research demonstrates significantly improved pain management in several pain conditions (e.g., rheumatoid arthritis, low-back pain, sports injuries); however, little is known about the effect of RSS with gamma-frequency sound stimulation on fibromyalgia. The use of RSS to treat fibromyalgia was first explored very recently and findings indicate that this treatment could be effective for individuals with fibromyalgia given that gamma-frequency sound stimulation indirectly stimulates neuronal coherence.

Aim: The present study aims to examine the effects of gamma frequency rhythmic sensory stimulation on fibromyalgia symptoms. Treatment effectiveness will be assessed by examining whether sensory stimulation will produce clinically meaningful changes in fibromyalgia symptom severity and whether treatment response will differ between the two treatment parameters.

Intervention: Fifty patients with a formal diagnosis of fibromyalgia were randomly assigned to two test groups. One group received vibrotactile stimulation from a continuous sine wave single-frequency stimulation (40 Hz) for 30 minutes, five days per week, over five weeks, concomitant with usual care. The second group completed the same treatment protocol but received different stimulation consisting of random and intermittent complex wave gamma-range vibrotactile stimulation. Measures of pain severity, fibromyalgia symptoms, sleep quality, and depression will be compared before and after treatment between the two groups.

The results of the present study will help to better understand the effectiveness of RSS for treatment of chronic pain disorders, such as fibromyalgia, and contribute to the development of future studies to investigate the mechanisms underlying clinical responses to rhythmic sensory stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of fibromyalgia conducted by the medical staff at Wasser Pain Management Centre;
* Ability to read and write English adequately;
* Have satisfactory hearing bilaterally (self-reported);
* Have the ability to operate the supplied device.

Exclusion Criteria:

* Acute and active inflammatory conditions (e.g., rheumatoid arthritis, osteoarthritis, autoimmune disease);
* Unstable medical or psychiatric illness;
* History of psychosis, epilepsy, seizures;
* Pregnancy or breast feeding;
* Hemorrhaging or active bleeding;
* Thrombosis, angina pectoris;
* Heart diseases, such as hypotension, arrhythmia, pacemaker;
* Substance abuse in the last year;
* Recently prolapsed vertebral disc;
* Recovering from a recent accident with back or neck injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change of Fibromyalgia symptoms and severity from baseline assessed by the Revised Fibromyalgia Impact Questionnaire (FIQ) at 6 weeks | Assessed at Week 0 (pre-intervention) and Week 6 (post-intervention)
  The FIQ is an assessment and evaluation instrument developed to measure fibromyalgia (FM) patient status, progress and outcomes, based on a 10 point scale.

SECONDARY OUTCOMES:
Change of sleep quality from baseline assessed by the Pittsburgh Sleep Quality Index (PSQI) at 6 weeks | Assessed at Week 0 (pre-intervention) and Week 6 (post-intervention)
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time.
Change of depression severity from baseline assessed by the Patient Health Questionnaire-9 (PHQ-9) at 6 weeks | Assessed at Week 0 (pre-intervention) and Week 6 (post-intervention)
  The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module.
Change in general quality of life from baseline assessed by the Quality of Life Enjoyment and Satisfaction questionnaire (Q-LES-Q-SF) at 6 weeks | Assessed at Week 0 (pre-intervention) and Week 6 (post-intervention)
  The Quality of Life Enjoyment and Satisfaction questionnaire is a generic, self-reported quality of life measure assessing the physical health, subjective feelings, leisure activities, social relationships, general activities, satisfaction with medications and life-satisfaction domains.
Change of pain severity from baseline assessed by Brief Pain Inventory - short form (BPI-SF) at 6 weeks | Assessed at Week 0 (pre-intervention) and Week 6 (post-intervention)
  BPI-SF is a 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning based on a 10 point scale.

OTHER OUTCOMES:
Patient Global Improvement Impression (PGI-I) | 6 weeks
  PGI-I is a global index that may be used to rate the response of a condition to a therapy.
Perceived treatment satisfaction assessed by a Modified version of the Glasgow Benefit Inventory | 6 weeks
  The Glasgow Benefit Inventory is a subjective post-interventional questionnaire especially developed to evaluate patient's perceived satisfaction with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Gordon, MD, Principal Investigator — MOUNT SINAI HOSPITAL; Lee Bartel, PhD, Study Director — University of Toronto
Locations (1):
- Wasser Pain Management Centre, Mount Sinai Hospital, Toronto, Ontario, Canada